CLINICAL TRIAL: NCT03439293
Title: A Phase 2, Open-Label Study of Ixazomib+Daratumumab+Dexamethasone (IDd) in Relapsed and/or Refractory Multiple Myeloma (RRMM)
Brief Title: A Study of Ixazomib+Daratumumab+Dexamethasone (IDd) in Relapsed and/or Refractory Multiple Myeloma (RRMM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16047; U1111-1202-6022 (Other: WHO); 2017-003977-32 (Registry Identifier: EudraCT)
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Multiple Myeloma
Keywords: Drug Therapy; Ixazomib; Daratumumab; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; daratumumab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ixazomib 4 mg + Daratumumab 16 mg/kg + Dexamethasone 20 mg (Experimental): Ixazomib, 4 mg, capsules, orally, on Days 1, 8 and 15 of each 28-day cycle along with daratumumab, 16 mg/kg, intravenously (IV), on Days 1, 8, 15 and 22 of Cycles 1 and 2, on Days 1 and 15 (every 2 weeks) for Cycles 3 to 6 and on Day 1 (every 4 weeks) for Cycle 7 and beyond along with dexamethasone, 20 mg, tablets, orally on Days 1, 2, 8, 9, 15, 16, 22 and 23 of each 28-day cycle until progressive disease (PD), unacceptable toxicity, or withdrawal of consent, or up to 5 years.
  Interventions: Drug: Ixazomib; Drug: Daratumumab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsule.
  Other Names: NINLARO
Drug: Daratumumab — Daratumumab IV infusion.
Drug: Dexamethasone — Dexamethasone tablets.

SUMMARY:
The purpose of this study is to evaluate the percentage of participants with a response of very good partial response (VGPR) or better to IDd treatment.

DETAILED DESCRIPTION:
The regimen being tested in this study is the combination of ixazomib, daratumumab, and dexamethasone. This study will look at the efficacy and safety of IDd in people who have RRMM.

The study will enroll approximately 60 Participants. Participants will be assigned to the treatment group:

• Ixazomib 4.0 mg + Daratumumab 16.0 mg/kg + Dexamethasone 20 mg

All participants will be asked to take Ixazomib on Days 1, 8 and 15 of each 28-day cycle plus Daratumumab on Days 1, 8, 15 and 22 of each 28-day cycle for Cycles 1 and 2, on Days 1 and 15 of each 28-day cycle for Cycles 3 through 6 and on Day 1 of each 28-day cycle for Cycle 7 and beyond plus Dexamethasone orally on Days 1, 2, 8, 9, 15, 16, 22 and 23 of each 28-day cycle.

This multi-center trial will be conducted in the United States, Czech Republic, France, Poland, Greece and the Netherlands. The overall time to participate in this study is approximately 5 years. Participants will make multiple visits to the clinic, and every 12 weeks after PD until death or termination of the study by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Have measurable disease by at least 1 of the following measurements:

   * serum M-protein >=1 gram per liter (g/dL) (>=10 g/L).
   * urine M-protein >=200 mg/24 hours.
2. Have documented evidence of PD on or after their last regimen as defined by IMWG criteria. All participants must have received between 1 to 3 prior therapies for MM (a prior therapy is defined as 2 or more cycles of therapy given as a treatment plan for MM [example, a single-agent or combination therapy or a sequence of planned treatments such as induction therapy followed by autologous stem cell transplant (SCT) and then consolidation and/or maintenance therapy]).
3. Have achieved a response (partial response (PR) or better) to at least 1 prior therapy.
4. Have an Eastern Cooperative Oncology Group (ECOG) score of 0, 1, or 2.
5. Must meet the following laboratory criteria:

   * Absolute neutrophil count (ANC) >=1000 per cubic millimeter (/mm^3).
   * Platelet count >=75,000/mm^3.
   * Total bilirubin less than or equal to (<=) 1.5*the upper limit of the normal range (ULN) (except for Gilbert syndrome: direct bilirubin <=2*ULN).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=3*ULN.
   * Calculated creatinine clearance >=50 mL/min.

Exclusion Criteria:

1. Have undergone prior allogenic bone marrow transplantation.
2. Have received prior ixazomib at any time or daratumumab or other anti-CD38 therapies, except as part of initial therapy if this was stopped to move on to SCT and the participant did not progress on anti-CD38 treatment.
3. Are refractory to bortezomib or carfilzomib at the last exposure before this study (defined as participants having PD while receiving bortezomib or carfilzomib therapy or within 60 days after ending bortezomib or carfilzomib therapy).
4. Are planning to undergo SCT prior to PD on this study (ie, these participants should not be enrolled in order to reduce disease burden prior to transplant).
5. Are receiving systemic treatment with strong Cytochrome P450 3A4 (CYP3A) inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital, St. John's wort) within 14 days before randomization.
6. Has received autologous SCT within 12 weeks before the date of study treatment.
7. With known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal. Note: FEV1 testing is required for participants suspected of having COPD and participants must be excluded if FEV1 is <50% of predicted normal.

   * Participants with Grade 2 or higher residual toxicities from prior therapy (including Grade 2 or higher peripheral neuropathy or any grade neuropathy with pain; excluding alopecia). This includes recovery from any major surgery. Note: Participants with planned surgical to be conducted under local anesthesia may participate. Kyphoplasty or vertebroplasty are not considered major surgery.
8. Has uncontrolled clinically significant cardiac disease, including myocardial infarction within 6 months before date of study entry or unstable or uncontrolled angina, congestive heart failure, New York Heart Association (NYHA) Class III-IV, uncontrolled cardiac arrhythmia (Grade 2 or higher).
9. With ongoing or active systemic infection requiring intravenous IV medical management ; participants with known human immunodeficiency virus- Ribonucleic acid (HIV-RNA) positivity; participants with hepatitis B virus (HBV) surface antigen or core antibody positivity; and participants with known hepatitis C virus-RNA positivity. Note: Participants who have positive hepatitis B core antibody can be enrolled but must have hepatitis B virus- deoxyribonucleic acid (DNA) negative. Participants who have positive hepatitis C antibody can be enrolled but must have hepatitis C virus-RNA negativity.

   Note: Participants who are already enrolled at the time of Amendment 02 should have local HBV testing performed as soon as possible for HBV surface antigen, e antigen, core antibody, and DNA. If any of these tests is positive, consult a physician with expertise in managing HBV for guidance regarding stopping daratumumab, starting HBV antiviral therapy, and remaining on study.
10. Diagnosed or treated for another malignancy within 2 years before randomization or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (28):
- United States (6):
  - Pacific Cancer Medical Center, Anaheim, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - SCRI - Florida Cancer Specialists - Panhandle, Tallahassee, Florida
  - Research Medical Center - Kansas City, Kansas City, Missouri
  - SCRI - Tennessee Oncology - Nashville - Centennial, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Czechia (5):
  - Fakultni Nemocnice Olomouc, Olomouc, Olomoucký kraj
  - Fakultni Nemocnice Kralovske Vinohrady, Prague, Prague
  - Fakultni Nemocnice Ostrava, Ostrava - Poruba, Severomoravsky KRAJ
  - Fakultni Nemocnice Brno, Brno
  - Onkologicka klinika Vseobecna fakultni nemocnice v Praze a 1, Prague
- France (4):
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Hopital Claude Huriez, Lille, Hauts-de-France
  - Hopital Hotel Dieu, Nantes, Pays de la Loire Region
  - Hopital Saint-Antoine, Paris, Île-de-France Region
- Greece (3):
  - Evaggelismos General Hospital, Athens, Attica
  - Alexandra General Hospital of Athens, Athens, Attica
  - University General Hospital of Patras Panagia I Voithia, Patras, Peloponnese
- Netherlands (5):
  - Vrije Universiteit Medisch Centrum, Amsterdam, North Holland
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Albert Schweitzer Ziekenhuis Dordwijk, Dordrecht, South Holland
  - Erasmus Medisch Centrum, Rotterdam, South Holland
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (5):
  - Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im. Ks. B. Markiewicza, Brzozów, Podkarpackie Voivodeship
  - Szpitale Pomorskie Spolka z ograniczona odpowiedzialnoscia, Gdynia, Pomeranian Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespol Szpitali Miejskich, Chorzów, Silesian Voivodeship
  - Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at investigative sites in Greece, the Czech Republic, the United States, Poland, France and the Netherlands from 13 March 2018 to 26 June 2023.
Pre-assignment Details: Participants with a diagnosis of relapsed and/or refractory multiple myeloma (RRMM) took part in the study to receive ixazomib + daratumumab + dexamethasone.
Period: Overall Study
Arm/Group | Ixazomib 4 mg + Daratumumab 16 mg/kg + Dexamethasone 20 mg
Started | 61
Response-evaluable Population (Response-evaluable population was defined as participants who received at least 1 dose of ixazomib, had measurable disease either during screening or before the first dose of study drug, and had a baseline and at least 1 postbaseline disease assessment.) | 59
Completed | 0
Not Completed | 61
Not completed — Death | 22
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 2
Not completed — Reason Not Specified | 28
Not completed — Missing | 1

BASELINE CHARACTERISTICS:
Population: Safety population included participants who received at least 1 dose of any study treatment regimen.
Arm/Group | Ixazomib 4 mg + Daratumumab 16 mg/kg + Dexamethasone 20 mg
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (7.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 53
  More than one race | 0
  Unknown or Not Reported | 5
Height [Mean (Standard Deviation); unit: centimeters (cm)] — Population: Number analyzed is the number of participants with data available for height at Baseline.
  centimeters (cm)
    number analyzed (Participants) | 60
    (all) | 166.8 (8.71)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 80.08 (17.625)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Very Good Partial Response (VGPR) or Better (Complete Response + VGPR)
Description: Response was assessed using International Myeloma Working Group (IMWG) Criteria. VGPR is defined as serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100 milligram (mg) per 24 hours. The percentage of participants were rounded off to the single decimal point.
Time Frame: Up to 5 years
Population: Response-evaluable population included participants who received at least 1 dose of ixazomib, had measurable disease during the screening period, and have at least 1 postbaseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib 4 mg + Daratumumab 16 mg/kg + Dexamethasone 20 mg
Number analyzed (Participants) | 59
percentage of participants | 32.2 [20.62 to 45.64]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as time from date of first dose of drug to date of first documentation of progressive disease (PD) or death from any cause, whichever occurs first. Participant without documentation of PD or death were censored at the date of last response assessment that is stable disease (SD) or better. PD is defined as increase of 25% of lowest response value in one or more of following criteria: serum M-component (absolute increase ≥0.5 g/dl); or urine M-component (absolute increase ≥200 mg/24-hour); difference between involved and uninvolved FLC levels (absolute increase >10 mg/dl); or bone marrow plasma cell percentage (absolute plasma cell percentage ≥10%); development of new/ increase in size of existing bone lesions or soft tissue plasmacytoma; or development of hypercalcemia that can be attributed solely to plasma cell proliferative disorder. SD is defined as not meeting criteria for other responses.
Time Frame: Up to 5 years
Population: Safety population included participants who received at least 1 dose of any study treatment regimen.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4 mg + Daratumumab 16 mg/kg + Dexamethasone 20 mg
Number analyzed (Participants) | 61
months | 16.8 [10.1 to 23.7]

3. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from the first dose of any study drug treatment to the date of the first documented PD. PD is defined as increase of 25% of lowest response value in one or more of following criteria: serum M-component (absolute increase ≥0.5 g/dl); or urine M-component (absolute increase ≥200 mg/24-hour); difference between involved and uninvolved FLC levels (absolute increase >10 mg/dl); or bone marrow plasma cell percentage (absolute plasma cell percentage ≥10%); development of new/ increase in size of existing bone lesions or soft tissue plasmacytoma; or development of hypercalcemia that can be attributed solely to plasma cell proliferative disorder.
Time Frame: Up to 5 years
Population: Safety population included participants who received at least 1 dose of any study treatment regimen.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4 mg + Daratumumab 16 mg/kg + Dexamethasone 20 mg
Number analyzed (Participants) | 61
months | 21.1 [10.2 to 27.9]

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of first dose of any study drug treatment to the date of death. Participant without documentation of death at the time of analysis will be censored at the last visit at which s/he was known to be alive.
Time Frame: Up to 5 years
Population: Safety population included participants who received at least 1 dose of any study treatment regimen.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4 mg + Daratumumab 16 mg/kg + Dexamethasone 20 mg
Number analyzed (Participants) | 61
months | NA [NA to NA] — Median, lower and upper limit of 95% confidence interval (CI) were not estimable due to low number of participants with events.

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as percentage of participants with complete response (CR), VGPR and partial response (PR). CR: Negative immunofixation of serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow; normal free light chain (FLC) ratio of 0.26-1.65; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or >=90% reduction in serum M-protein + urine M-protein level <100 mg/24 hours; and PR: >=50% reduction of serum M protein and reduction in 24-hour urinary M protein by >=90%/to <200 mg/24 hours; In addition, if present at baseline, >=50% reduction in size of soft tissue plasmacytomas; no known evidence of progressive/new bone lesions. The percentage of participants were rounded off to the single decimal point.
Time Frame: Up to 5 years
Population: Response-evaluable population included participants who received at least 1 dose of ixazomib, had measurable disease during the screening period, and had at least 1 postbaseline disease assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Ixazomib 4 mg + Daratumumab 16 mg/kg + Dexamethasone 20 mg
Number analyzed (Participants) | 59
percentage of participants | 66.1

6. Secondary Outcome: Time To Response (TTR)
Description: TTR is defined as the time from first dose of any study drug treatment to the date of first documentation of PR or better. PR is defined as >=50% reduction of serum M protein and reduction in 24-hour urinary M protein by >=90%/to <200 mg/24 hours; In addition, if present at baseline, >=50% reduction in size of soft tissue plasmacytomas; no known evidence of progressive/new bone lesions.
Time Frame: Up to 5 years
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4 mg + Daratumumab 16 mg/kg + Dexamethasone 20 mg
Number analyzed (Participants) | 59
months | 2.7 [1.9 to 5.8]

7. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the date of first documentation of PR or better to the date of the first documented PD among participants who responded to the treatment.
Time Frame: Up to 5 years
Population: Response-evaluable population included participants who received at least 1 dose of ixazomib, had measurable disease during the screening period, and had at least 1 postbaseline disease assessment. The data is reported for the responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4 mg + Daratumumab 16 mg/kg + Dexamethasone 20 mg
Number analyzed (Participants) | 39
months | 24.0 [15.9 to NA] — Upper limit of 95% CI was not estimable due to low number of responders with events.

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Safety population included participants who received at least 1 dose of any study treatment regimen.
Arm/Group | Ixazomib 4 mg + Daratumumab 16 mg/kg + Dexamethasone 20 mg
All-Cause Mortality (participants affected / at risk) | 22/61
Serious Adverse Events (participants affected / at risk) | 28/61
Other Adverse Events (participants affected / at risk) | 58/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib 4 mg + Daratumumab 16 mg/kg + Dexamethasone 20 mg (N=61)
Acute kidney injury (Renal and urinary disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bronchitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 2
COVID-19 pneumonia (Infections and infestations) | 3
Cardiovascular disorder (Cardiac disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Gastroenteritis (Infections and infestations) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Influenza B virus test positive (Investigations) | 1
Loss of consciousness (Nervous system disorders) | 1
Monoclonal immunoglobulin present (Investigations) | 1
Necrotising fasciitis (Infections and infestations) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Pneumonia herpes viral (Infections and infestations) | 1
Pneumonia legionella (Infections and infestations) | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1
Pseudomonal bacteraemia (Infections and infestations) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Spinal cord compression (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Sudden death (General disorders) | 1
Syncope (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Vestibular disorder (Ear and labyrinth disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib 4 mg + Daratumumab 16 mg/kg + Dexamethasone 20 mg (N=61)
Abdominal pain upper (Gastrointestinal disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Asthenia (General disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Bronchitis (Infections and infestations) | 8
Cataract (Eye disorders) | 6
Constipation (Gastrointestinal disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 26
Dizziness (Nervous system disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Fall (Injury, poisoning and procedural complications) | 6
Fatigue (General disorders) | 15
Headache (Nervous system disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 7
Hypoaesthesia (Nervous system disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 6
Infusion related reaction (Injury, poisoning and procedural complications) | 4
Insomnia (Psychiatric disorders) | 9
Leukopenia (Blood and lymphatic system disorders) | 5
Lower respiratory tract infection (Infections and infestations) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Nasopharyngitis (Infections and infestations) | 5
Nausea (Gastrointestinal disorders) | 13
Neuropathy peripheral (Nervous system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 4
Oedema peripheral (General disorders) | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 6
Peripheral swelling (General disorders) | 4
Pneumonia (Infections and infestations) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6
Pyrexia (General disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Somnolence (Nervous system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 16
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 6
Vertigo (Ear and labyrinth disorders) | 4
Vomiting (Gastrointestinal disorders) | 6
White blood cell count decreased (Investigations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT03439293/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT03439293/SAP_001.pdf